CLINICAL TRIAL: NCT02651792
Title: Ketamine-propofol Versus Pethidine-propofol for Sedating Patients Undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP)
Brief Title: Ketamine- Propofol Versus Pethidine- Propofol in ERCP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, khaled salah mohamed, lecturer of anaesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ketfol versus pethidine
Record Dates: First submitted 2015-11-29; First posted 2016-01-11 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Sedation in ERCP
Keywords: ketamine; propofol; pethidine; ERCP; endoscopist

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- ketamine- propofol (Active Comparator): IV Ketamine 1mg/kg + Propofol 1.2 mg/kg will be given for sedation.
  Interventions: Drug: ketamine- propofol
- pethidine- propofol (Active Comparator): 1.1 mg x kg(-1) pethidine + 1.2 mg x kg(-1) propofol for sedation induction
  Interventions: Drug: pethidine- propofol

INTERVENTIONS:
Drug: ketamine- propofol — 1 mg x kg(-1) ketamine + 1.2 mg x kg(-1) propofol.
  Other Names: N01AX03 - Propofol
  Arms: ketamine- propofol
Drug: pethidine- propofol — 1.1 mg x kg(-1) pethidine + 1.2 mg x kg(-1) propofol for sedation induction
  Other Names: meperidine - Propofol
  Arms: pethidine- propofol

SUMMARY:
The investigators aim to investigate the differences between ketamine propofol and pethidine propofol during ERCP in respect to endoscopist satisfaction.

DETAILED DESCRIPTION:
The investigators aim to investigate the differences between ketamine propofol and pethidine propofol during ERCP in respect to endoscopist satisfaction, amount of propofol consumption Any desaturation or apnea will be recorded when the oxygen saturation (SpO2) dropped to <90% , time for recovery ,post-operative nausea and vomiting, hallucinations and Ramsey sedation scores of all patients will be recorded perioperatively. The Aldrete score was used to measure recovery from anesthesia at 5 and 10 min after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* both gender
* age between 18-70

Exclusion Criteria:

* pregnant patients.
* morbid obesity.
* chronic obstructive pulmonary disease.
* complicated airway.
* American society of anesthesia (ASA) physical classification IV-V.
* history of allergy or contraindications to the drugs used in the study
* emergency need for ERCP.
* those whose informed consent could not be signed.
* those with possible complex ERCP.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
endoscopist satisfaction using 5 step scale (5= optimal condition; 1= poor condition) | Immediately after procedure.

OTHER OUTCOMES:
amount of propofol consumed during procedure | Immediately after procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa S Abbas, MD, Study Chair — Assiut University
Locations (1):
- Al Rajhy liver hospital, Asyut, Egypt